CLINICAL TRIAL: NCT03135145
Title: Post-operative Use of Lite Run in a Pediatric Population With Cerebral Palsy
Brief Title: Post-operative Lite Run Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: Lite Run Inc. (Industry)
Responsible Party: Principal Investigator, Joyce Trost, Manager of Research Administration, Gillette Children's Specialty Healthcare
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: LiteRun-001
Record Dates: First submitted 2017-03-22; First posted 2017-05-01 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy; Neurologic Disorder; Chromosome Abnormality; Spina Bifida
Keywords: Single Event Multilevel Lower Extremity Orthopedic Surgery (SEMLS); Physical Therapy; Gait Training; Functional Walking; Selective Dorsal Rhizotomy (SDR)
MeSH Terms: conditions — Cerebral Palsy; Nervous System Diseases; Chromosome Aberrations; Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: This is a single group repeated measures cross-over design. The study will include 4 sessions for each participant, with 2 sessions conducted using the Lite Run and 2 sessions conducted using the method of choice of the therapist (Usual Treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Lite Run Gait Trainer (Active Comparator): Participants will be using the Lite Run Gait Trainer to assist them in weightbearing and walking after SDR or SEMLS surgery.
  Interventions: Device: Lite Run Gait Trainer
- Usual Treatments (Placebo Comparator): Participants will be using current treatments used in clinical practice to assist them in weightbearing and walking after SDR or SEMLS surgery.
  Interventions: Other: Usual Treatments

INTERVENTIONS:
Device: Lite Run Gait Trainer — Lite Run is a new system for the treatment of patients with gait and balance difficulties that uses differential air pressure inside a lower body suit to reduce up to 50 percent of a patient's body weight. The suit is similar to a pair of pants in appearance and is as easy to don and doff as a pair of pants. The suit uses technology like astronaut spacesuits to achieve comfort and flexibility while providing a unique "unweighting" effect that facilitates patient ambulation from sitting through taking steps. The suit is used in conjunction with the Lite Run Gait Trainer, which provides air pressure to the suit and support for the patient.
  Other Names: Lite Run; DHF No: 55-0001, 55-0002 & 55-0003
  Arms: Lite Run Gait Trainer
Other: Usual Treatments — The usual clinical treatments (standard of care treatments) will be used to assist patients in weightbearing and walking.
  Arms: Usual Treatments

SUMMARY:
Lite Run is a new assistive device that may have FDA listing as a Class I device by mid 2017 based on clinical testing of adults, independent agency testing and in-house evaluations.

This will be a combined study with multiple purposes with respect to the evaluation of its use with the post-operative pediatric population. A first purpose is to verify safety and feasibility of the device on pediatric patients. A second purpose is to statistically test the effectiveness of Lite Run to decrease physical burden on the therapist during post-operative gait training for children and adolescents with cerebral palsy as compared to current methods of body weight-supported gait training. A third purpose is to measure and qualitatively evaluate the effectiveness of the device on patient outcomes and improving patient and therapist satisfaction.

DETAILED DESCRIPTION:
Background Cerebral palsy (CP) refers to a group of disorders affecting movement and is attributable to a non-progressive injury to the developing brain. CP is the most common cause of physical disability in childhood with a prevalence of 3.1 - 3.6 per 1000 births. At this prevalence, we estimate that over 300,000 children under 21 in the US have CP. Children with CP have a variety of neuro-motor impairments including muscle weakness and abnormal muscle tone that leads to progressive musculoskeletal impairments over time. These children experience discomfort and limitations in functional mobility such as walking (ambulation) that severely impact their quality of life. Surgical intervention is often used to improve ambulation quality and quantity for children with cerebral palsy anytime from childhood into adulthood. Depending on treatment goals, it is not unusual for an individual with cerebral palsy to undergo surgery involving muscles, tendons, bones or nerves of the feet, ankles, legs or hips. Two common surgical interventions for ambulatory children with cerebral palsy include single event multilevel orthopedic surgery to correct muscle lengths and bone alignment, and selective dorsal rhizotomy to decrease spasticity. Post-operative treatment course varies depending on the child's condition, pre-operative functional level, and specific surgical intervention selected to improve their particular deficiencies. Post-orthopedic surgery, children may be non-weight-bearing for 2-6 weeks. After selective dorsal rhizotomy, patients exhibit surgical site instability and significant trunk and leg weakness. They are non-weight-bearing for 2-4 weeks post-surgically, and may begin to stand and walk once cleared by the physician.

When beginning mobility training after orthopedic or selective dorsal rhizotomy surgery, children typically demonstrate significant weakness and can experience fear, pain and anxiety as they begin to move. One aspect of mobility that is a significant milestone for children post-surgically is getting back up and walking. The process to get back up and walk is facilitated by physical therapists and is termed "gait training" which includes the components of moving from sit to stand, bearing weight through the lower limbs, taking steps, and returning to a sitting position. Body weight-supported gait training is often used in therapy for adults and children to ease the transition from non-weight-bearing back to being able to walk at their previous level of gait function. Support during this transition may be provided by a physical therapist using a gait belt, a harness system attached to an overhead track or device to support body weight, or other assistive devices. Current body weight support systems for gait training are not optimal. Also there are reports in the literature of difficulties with harness discomfort and donning and doffing. An unpublished survey of twelve physical therapists was conducted by a University of Minnesota PT student who was able to identify 20 deficiencies in available devices for body weight supported gait training. More than 50% of the therapists cited the following sub-optimal aspects from their experiences:

* Therapist providing majority of the body weight support when using a gait belt takes away from therapeutic touch for gait therapy
* Current harness devices cannot adjust the percent of how much support the device gives
* There is not sufficient therapeutic evidence for the efficacy of current body weight support devices
* Current harness devices do not feel like they will help us prevent injury.
* Current body weight support devices only work in limited applications

Using physical therapist support for gait training without a body weight support device can require multiple people to assist, result in fatigue, and has the potential of injury for the therapist. In a survey of physical therapists working in rehabilitation facilities, 67% reported musculoskeletal pain or discomfort within the past year. Half reported that patient repositioning (49%) and gait training (47%) also caused or contributed to their pain. Another study reports survey results of over 1,000 occupational and physical therapists. The survey indicated that functional activities such as gait training and settings such as pediatric rehabilitation were associated with injury. An ergonomic analysis of physical therapists working in rehabilitation concluded that physical therapists are at high risk for work related musculoskeletal injuries while performing sit-to-stand transfers and overground gait training.

To improve gait training therapy for both therapist and patient and to reduce a therapist's need to lift and support the body weight of a patient, Lite Run Inc. has developed the Lite Run Gait Trainer (Lite Run). Lite Run is a new system for the treatment of patients with gait and balance difficulties that uses differential air pressure inside a specially designed lower body suit to effectively reduce up to 50 percent of a patient's body weight. The suit is similar to a pair of pants in appearance and is as easy to don and doff as a pair of pants. The suit uses technology like astronaut spacesuits to achieve comfort and flexibility while providing a unique "unweighting" effect that facilitates patient ambulation from sitting through taking steps. The suit is used in conjunction with the Lite Run Gait Trainer, which provides air pressure to the suit and support for the patient.

Lite Run features include: (1) control for the amount of body weight support (up to 50% of the patient's weight), (2) electro-mechanical and pneumatic controls for providing assistance in transferring the patient from sitting to standing and ambulation, (3) an open design that permits access to a patient's body and legs by the therapist, (4) a compact profile that provides easy maneuverability, and (5) a "base spread" function that permits positioning close to a patient when seated in a wheelchair, bed or therapy table.

Together, these features provide safety and stability for the patient and reduced physical burden on the therapist while improving the gait training experience and potentially preventing patient or therapist injury. The system also frees the therapist to focus on skilled therapeutic activities because the patient is secure in the system.

Lite Run conducted a product demonstration and pediatric needs survey for six physical therapists at Gillette Children's Specialty Healthcare. Current support devices used for training include overhead harness supports, robotic systems, and harness gait trainers. Therapists indicated that current devices can be uncomfortable, cause patients to "hang" on the support, and limit natural motion during sit-to-stand and walking. Gait trainers and walking devices provide trunk and pelvic support using a seat or harness, and are used with a treadmill which can be both uncomfortable and scary for children right out of surgery.

Lite Run may have FDA listing as a Class I device by mid 2017 based on adult clinical feasibility testing, and completion of independent agency testing and in-house evaluations. A clinical safety and feasibility trial for adult patients was performed at the Rehabilitation Center at North Memorial Medical Center, Robbinsdale, MN with 18 adults with a range of neurological conditions.

Adult physical therapists participating in this trial have indicated the following:

* Lite Run is comfortable. Harnesses at the groin are uncomfortable for many patients. Lite Run has the potential to decrease pain, and improve security, support, compression, adjustability, and flexibility in combination with support. It provides improved mobility during sit-to-stand. The device may allow the patient to get back up walking sooner after surgery than if they were using another device.
* It is easy for therapists to use. Pants donning time is less than 5 minutes, and requires two quick attach points to engage the patient into the device. It is easily adjustable.
* It decreases the burden on the therapist. Because the device supports the patient's body weight, therapists hands are free to provide cuing and facilitation rather than physical support. It could prevent therapist injury particularly to the back. It is fall proof.
* The device is able to quantify the amount of support provided.

The results of this study indicated that there were no adverse events or safety issues from using the system on adults. In addition to safety and feasibility testing, the following user design requirements were tested: time to don liner and pants, transfer-in time, therapist's access to patient, patient's arm mobility, hindrance of patient's stride, patient directed steerability, brake stability, overall stability, sit-to-stand functionality, wheelchair compatibility, sit-to-stand sufficiency, odometer acceptability, ease of use, and the physical effort required by the PT. After training, all therapists were all able to operate the Lite Run safely and independently. The device allowed them to use their hands to provide skilled therapeutic maneuvers, as the device provided stability and patient unweighting. The study demonstrated that the Lite Run is a safe system and shows potential for pediatric application to improve the rehabilitation experience and outcomes. Therefore, continued investigation regarding the feasibility of using the device in a post-operative pediatric population using pediatric sized lower body pressure suits is warranted.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cerebral palsy, neurologic syndrome, chromosomal abnormalities, spina bifida, or other neurological disorders
* age 4-17
* recent single event multilevel lower extremity orthopedic surgery or selective dorsal rhizotomy
* referred for physical therapy for mobility/gait training to regain functional walking and ambulation

Exclusion Criteria:

* Gross Motor Function Classification System levels I (walk and run in the community with only limitations in balance, coordination and speed) and V (use wheelchair to maintain sitting and for whole body mobility) prior to surgical intervention
* Subjects who are too large or too small to fit within the current Lite Run pants/prototype. The minimum patient weight is 50 lbs. The maximum patient weight is 350 lbs.
* Subjects that do not have clearance for full weight-bearing at the first treatment session

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed by CTCAE v, 4. | Through study completion, up to 60 days
  Adverse events will be tracked for each subject enrolled in the study.
Number of Pass or Fail grades for setting up the Lite Run device | Through study completion, up to 60 days
  This measure will look at how easy Lite Run is to set up with a Pass or Fail grade by a trained Observer.
Reduction of physical assistance by study Physical Therapists as assessed by the ordinal scale for the Walk item of the WeeFim II ® Locomotion subscale | Through study completion, up to 60 days
  This measure will look at whether use of the Lite Run device will decrease the physical assistance needed for ambulation compared to standard of care treatments.

SECONDARY OUTCOMES:
Reduction of physical assistance for sit-to-stand mobility for participants assessed by the ordinal scale 1-6 for the Transfer: Chair item of the WeeFIM II® Transfer subscale | Through study completion, up to 60 days
  The will measure the amount of physical assistance needed for the sit-to-stand motion during physical therapy.
Increased duration of therapeutic weight-bearing activities in minutes | Through study completion, up to 60 days
  A trained observer will document the number of minutes spent doing weightbearing activities during study visits to see if there is an increase when using the Lite Run device.
Reduction of Pain during physical therapy for Non-Verbal children assessed by the Non-communicating Children's Pain Check List - Postoperative Version | Through study completion, up to 60 days
  Pain during study Visits will be assessed with the Non-communicating Children's Pain Check List - Postoperative Version for any children who are non-verbal. It is hypothesized that pain will be reduced when the Lite Run device is used during therapy.
Reduction of Pain during physical therapy for Children | Through study completion, up to 60 days
  Pain during the study Visits will be assessed with the Visual Analog Pain Scale. It is hypothesized that pain will be reduced when using the Lite Run device during therapy.
Reduction of Anxiety levels during therapy for children ages 8 to 17 years will be assessed with the Visual Analog Anxiety Scale . | Through study completion, up to 60 days
  Anxiety will be measured at each study visit with the Visual Analog Anxiety Scale. It is hypothesized that anxiety will be reduced when using the Lite Run device during therapy.
Reduction of Anxiety levels during therapy for children ages 4-7 years will be assess with the Children's Fear Scale "Scared". | Through study completion, up to 60 days
  Anxiety will be measured at each study visit with the Children's Fear Scale "Scared". It is hypothesized that anxiety will be reduced when using the Lite Run device during therapy.
Participant Satisfaction will be measured after each therapy visit with the QUEST Version 2.0 will be used, focusing on the first eight questions. | Through study completion, up to 60 days
  Participant satisfaction with their therapy will be measured with the QUEST Version 2.0 will be used, focusing on the first eight questions. We hypothesize that participants will have a higher satisfaction score when the Lite Run device is used at their therapy visit
Therapist Satisfaction will be measured after each therapy visit with the QUEST Version 2.0 will be used, focusing on the first eight questions. | Through study completion, up to 60 days
  Therapist satisfaction with the participants therapy will be measured using the QUEST Version 2.0 will be used, focusing on the first eight questions. We hypothesize that therapists will have a higher satisfaction score when the Lite Run device is used during the therapy visit.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Trost, PT, Principal Investigator — Gillette Children's Specialty Healthcare; John Hauck, Principal Investigator — Lite Run Inc.; Doug Johnson, Principal Investigator — Lite Run Inc.
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaslund MK, Moe-Nilssen R. Treadmill walking with body weight support effect of treadmill, harness and body weight support systems. Gait Posture. 2008 Aug;28(2):303-8. doi: 10.1016/j.gaitpost.2008.01.011. Epub 2008 Mar 17. PMID 18343664
- [Background] Azaula M, Msall ME, Buck G, Tremont MR, Wilczenski F, Rogers BT. Measuring functional status and family support in older school-aged children with cerebral palsy: comparison of three instruments. Arch Phys Med Rehabil. 2000 Mar;81(3):307-11. doi: 10.1016/s0003-9993(00)90076-5. PMID 10724075
- [Background] Bell KJ, Ounpuu S, DeLuca PA, Romness MJ. Natural progression of gait in children with cerebral palsy. J Pediatr Orthop. 2002 Sep-Oct;22(5):677-82. PMID 12198474
- [Background] Breau LM, Finley GA, McGrath PJ, Camfield CS. Validation of the Non-communicating Children's Pain Checklist-Postoperative Version. Anesthesiology. 2002 Mar;96(3):528-35. doi: 10.1097/00000542-200203000-00004. PMID 11873023
- [Background] Christensen D, Van Naarden Braun K, Doernberg NS, Maenner MJ, Arneson CL, Durkin MS, Benedict RE, Kirby RS, Wingate MS, Fitzgerald R, Yeargin-Allsopp M. Prevalence of cerebral palsy, co-occurring autism spectrum disorders, and motor functioning - Autism and Developmental Disabilities Monitoring Network, USA, 2008. Dev Med Child Neurol. 2014 Jan;56(1):59-65. doi: 10.1111/dmcn.12268. Epub 2013 Oct 1. PMID 24117446
- [Background] Darragh AR, Campo M, King P. Work-related activities associated with injury in occupational and physical therapists. Work. 2012;42(3):373-84. doi: 10.3233/WOR-2012-1430. PMID 22523031
- [Background] Han B, Enas NH, McEntegart D. Randomization by minimization for unbalanced treatment allocation. Stat Med. 2009 Nov 30;28(27):3329-46. doi: 10.1002/sim.3710. PMID 19739238
- [Background] Hanna SE, Rosenbaum PL, Bartlett DJ, Palisano RJ, Walter SD, Avery L, Russell DJ. Stability and decline in gross motor function among children and youth with cerebral palsy aged 2 to 21 years. Dev Med Child Neurol. 2009 Apr;51(4):295-302. doi: 10.1111/j.1469-8749.2008.03196.x. PMID 19391185
- [Background] Johnson DC, Damiano DL, Abel MF. The evolution of gait in childhood and adolescent cerebral palsy. J Pediatr Orthop. 1997 May-Jun;17(3):392-6. PMID 9150031
- [Background] McKinley S, Coote K, Stein-Parbury J. Development and testing of a Faces Scale for the assessment of anxiety in critically ill patients. J Adv Nurs. 2003 Jan;41(1):73-9. doi: 10.1046/j.1365-2648.2003.02508.x. PMID 12519290